CLINICAL TRIAL: NCT05025709
Title: Bronchospasm During Anesthetic Induction: Study of Clinical Characteristics and Treatments Administered According to Etiology
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, MOUTON-FAIVRE Claudie, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI277
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Bronchospasm
Keywords: bronchial spasm; general anaesthesia; allergy; anaphylaxis
MeSH Terms: conditions — Bronchial Spasm; Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchospasm during anaesthesia is a rare but potentially life-threatening event. They are classically part of IgE-dependent anaphylaxis but can also occur as an independent clinical entity, triggered by inflammatory factors such as smoking, chronic bronchitis, asthma, overweight and mechanical factors such as tracheal intubation.

The etiological diagnosis is currently established during an allergy-anaesthesia consultation after skin testing for drugs used for induction of anaesthesia and antibiotic therapy when it is attributable.

The aim of this study was to determine the characteristics that differ between 2 groups: isolated non-allergic bronchospasm and bronchospasm as part of an immediate allergic hypersensitivity reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the allergy consultation for investigation of an immediate hypersensitivity reaction, involving a bronchospasm explicitly identified by the anaesthetist, which occurred during an anaesthetic procedure.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients included were those referred to the allergy consultation (dermato-allergology department of the Nancy University Hospital), over a period from October 2017 to March 2021, for investigation of an immediate hypersensitivity reaction, involving a bronchospasm explicitly identified by the anaesthetist, which occurred during an anaesthetic procedure. There were no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical reactions | Baseline (J0)
  To show that clinical reactions presented by patients with non-allergic bronchospasm are different from those presented with allergic bronchospasm (Presence or absence of associated signs such as hypotension, heart rate variation, skin signs, desaturation, EtCO2 variation).
Treatments provided | Baseline (J0)
  To determine whether the treatments provided to patients with non-allergic bronchospasm are different from those provided to patients with allergic bronchospasm.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermato-allergology department of the Nancy University Hospital, Nancy, France